CLINICAL TRIAL: NCT02294591
Title: NACOS - The Effect of N-acetylcystein for Depressive Symptoms in Patients Suffering From Bipolar Depression - A Double Blind Randomized Placebo-controlled Trial With Follow up
Brief Title: NACOS - The Effect of N-acetylcystein for Depressive Symptoms in Patients Suffering From Bipolar Depression
Acronym: NACOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Syddanmark (Other)
Responsible Party: Principal Investigator, Connie Thuree Nielsen, consultant, MD, ph.d, Consultant, MD, Ph.D, Region Syddanmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35664; 2012-004483-22 (EudraCT Number)
Record Dates: First submitted 2014-11-06; First posted 2014-11-19 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Depression; Acetylcystein; Oxidative Stress; Urine
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC group (Active Comparator): Receiving N-acetylcysteine as add-on treatment
  Interventions: Drug: N-acetylcysteine
- Placebo group (Placebo Comparator): Receiving placebo as add-on treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Add-on treatment of NAC
  Other Names: NAC
  Arms: NAC group
Drug: Placebo — Add-on treatment of placebo
  Arms: Placebo group

SUMMARY:
This trial investigate add-on treatment with 3 g NAC vs. placebo in 20 weeks in patients suffering from bipolar depression. The primary outcome is MADRS-score, and the secondary outcomes are other psychometric evaluations oxidative stress biomarkers in urine.

DETAILED DESCRIPTION:
Bipolar depression can be extremely invalidating because of the depressive symptoms that results in decreased social functioning which reduces the quality of life. Bipolar depression is associated with three times longer duration of disorder period compared to mania. This emphasizes the importance of optimal treatment opportunities for this particular group.

Psychological treatments are often based on effective maintenance therapy, with limited evidence of acute bipolar depression. The effect of lithium in the acute phase of depression is low, and the use of valproate is still unclear in bipolar depression. Lamotrigine and other antipsychotics, has some efficacy in bipolar depression but have considerable tolerance issue. The most effective treatment is quetiapine and quetiapine XR, but this treatment is associated with side effects such as sedation, weight gain and dyslipidemia.

Individuals suffering from bipolar depression has a recognisable dysregulated oxidative mechanisms. Evidence indicates that GSH, which is the central antioxidant in brain are vulnerable to degradation. However, N-acetylcystine (NAC) improves the L-cysteine supply and leads to increase GSH in the brain.

A clinical randomized controlled study with 75 patients, showed a significant decreases in the primary outcome measure (MADRS-score) compared to the control group. Furthermore, were the general health status and function improved in NAC group.

This double-blinded randomized placebo controlled trial is conducted, to demonstrate the efficacy of NAC on depressive symptoms in patients suffering from bipolar depression, and examine the effect of add-on treatment of NAC on the level of oxidative stress, quality of life and functioning.

In total 87 participants will be included and recruited from The Mental Health Service from Region of Southern Denmark, to ensure sufficient participants in the study.

The trial will run for a 24 weeks period for each participant. Participants in the study will be randomized to either NAC and standard treatment, or placebo and standard treatment for 20 weeks, followed by a 4-week follow-up period.

This trial is the first of its kind, analysing the level of oxidative stress in both blood and urine samples among people suffering from bipolar depression, to examine the add-on effect of NAC treatment.

The study receive academic and scientific advice from Ramus W. Licht, professor, ph.d, and clinical advice from Henrik E. Poulsen, professor, dr.med. This is two international professors in respectively bipolar disorder and oxidative stress. Furthermore, there is an international corporation and support from professor Michael Berk and dr. Olivia Dean from Deakin University, Australia, which have performed the previously trials concerning NAC treatment and bipolar depression.

The study medication has low side effects and low cost, both advantages, which are desirable for especially this vulnerable group of people. This trial may contribute to optimal treatment opportunities for people suffering from bipolar depression, and possibly other psychiatric patients as well.

ELIGIBILITY:
Inclusion Criteria:

Patients that meet the DSM-5 criteria of bipolar disorder type 1 or 2 (296-41-296.56 or 296.89) with at least one documented illness episode in the past six months, have had depressive symptoms at least 4 weeks before inclusion, MADRS ≥ 18 at baseline, have been sick at least 4 weeks, between 18-64 years, fertile women with a negative pregnant test at baseline, turtle women using safe contraception in the study period, and patients who have given informed consent.

Exclusion Criteria:

Pregnant women, patients wishing pregnancy during the frame of the study, current suicidality, patients that have an intake of more than 500 mg NAC, 200 μm selenium, or 500 IU of vitamin E every day is excluded. Patients who are hypersensitive to histamine, patients who have had ECT-treatment within the last 4 weeks. Patients with recent bleeding in respiratory, asthma, epilepsy or allergy towards NAC. People who cannot speak or understand the Danish language, or have not give or withdrawn informed consent. If patients change diagnosis during the study, and the primary diagnosis is not bipolar affective disorder is the participant excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The total score of MADRS | Change from baseline MADRS-score at 20 weeks

SECONDARY OUTCOMES:
The total score of MES | Change from baseline MES-score at 20 weeks
The total score of WHO-5 | Change from baseline WHO-5-score at 20 weeks
The total score of GAF-S | Change from baseline GAF-S-score at 20 weeks
The total score of GAF-F | Change from baseline GAF-F-score at 20 weeks
The total score of YMRS | Change from baseline YMRS-score at 20 weeks
The measurement of oxidative stress in biological material (urine) | Change from baseline oxidative stress measurement at 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Connie T. Nielsen, Ph.D, Principal Investigator — Mental Health Service, Esbjerg
Locations (1):
- Mental Health Services Esbjerg, Esbjerg, Denmark

REFERENCES:
- [Derived] Ellegaard PK, Licht RW, Poulsen HE, Nielsen RE, Berk M, Dean OM, Mohebbi M, Nielsen CT. Add-on treatment with N-acetylcysteine for bipolar depression: a 24-week randomized double-blind parallel group placebo-controlled multicentre trial (NACOS-study protocol). Int J Bipolar Disord. 2018 Apr 5;6(1):11. doi: 10.1186/s40345-018-0117-9. PMID 29619634